CLINICAL TRIAL: NCT03295214
Title: A Prospective Clinical Trial Evaluating the Post-Operative Analgesic Effects of Acetaminophen Given Per Os and Intravenous
Brief Title: Acetaminophen Given Per Os and Intravenous in Sinus Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Luliu Fat, Principal Investigator, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1098410
Record Dates: First submitted 2017-09-21; First posted 2017-09-27 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Acetaminophen
Keywords: Acetaminophen; Functional Endoscopic Sinus Surgery
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetaminophen 975mg Per Os (Active Comparator): 975mg of Acetaminophen given by mouth
  Interventions: Drug: Acetaminophen
- Acetaminophen 1000mg Intravenous (Active Comparator): 1000mg of Acetaminophen given intravenously
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen given for pain relief

SUMMARY:
The primary objective of this study is to investigate the Visual Analog Score (VAS) for pain within the post-operative setting and determine if there is a statistically significant difference between the VAS for PO or IV acetaminophen. It is expected that in doing so the investigators can produce the maximal amount of pain relief after surgery while making conscientious monetary decisions.

DETAILED DESCRIPTION:
Functional Endoscopic Sinus Surgery (FESS) is one of the most common Ear Nose and Throat Surgeries done in the United States annually. This procedure can vary from intense to moderate pain and as such it is difficult to properly gauge and treat postoperative pain in these patients. Commonly used in these cases, opioid drugs are given to provide adequate analgesia, however higher opioid usage is observed to cause increased Post-Anesthesia Care Unit (PACU) stays, respiratory complications and Postoperative Nausea and Vomiting (PONV). Acetaminophen is commonly used as an adjunct in these circumstances because of its opioid sparing properties.

Acetaminophen is a synthetic nonopioid p-aminophenol derivative available over the counter. Its properties include analgesic and antipyretic qualities and it is listed on the world health organization's list of essential medicines. The potential risks include liver damage, skin reactions and drug interactions when used with blood thinners at high doses. Acetaminophen has been extensively researched, in vitro and in vivo studies have found the drug to be safe when used at proper doses. Recently intravenous use of acetaminophen has gained popularity due to ease of use and ability to be given intraoperatively. This form of acetaminophen, although convenient, is around sixty two times the cost of oral acetaminophen. Due to this increased cost it is imperative that the investigators compare the two routes of administration in order to determine if the additional cost is justified.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate
* Undergoing FESS surgery at Massachusetts Eye and Ear (MEE)
* Over the age of 18 during time of surgery
* Weighing over 50kg

Exclusion Criteria:

* Severe hepatic impairment or active liver disease
* Known hypersensitivity to acetaminophen or to any excipients in the intravenous formulation
* chronic opioid use
* chronic pain
* alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
VAS for pain | 0-1 hour
  First VAS pain score applied

SECONDARY OUTCOMES:
Opioid Use | 24 hours
  Postoperative opioid consumption for pain control
Time in PACU | 3-5 hours
  Time required to be admitted and discharged home
VAS for pain | 1-2 hours
  Second VAS pain score applied
VAS for pain | 2-3 hours
  Third VAS pain score applied
VAS for pain | 24 hours
  Last VAS pain score applied
PONV | 24 hours
  Incidence of PONV

CONTACTS AND LOCATIONS:
Overall Officials: Iuliu Fat, MD, Principal Investigator — MEEI
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carroll NV, Miederhoff PA, Cox FM, Hirsch JD. Costs incurred by outpatient surgical centers in managing postoperative nausea and vomiting. J Clin Anesth. 1994 Sep-Oct;6(5):364-9. doi: 10.1016/s0952-8180(05)80004-2. PMID 7986507
- [Background] DeLoach LJ, Higgins MS, Caplan AB, Stiff JL. The visual analog scale in the immediate postoperative period: intrasubject variability and correlation with a numeric scale. Anesth Analg. 1998 Jan;86(1):102-6. doi: 10.1097/00000539-199801000-00020. PMID 9428860
- [Background] Fenlon S, Collyer J, Giles J, Bidd H, Lees M, Nicholson J, Dulai R, Hankins M, Edelman N. Oral vs intravenous paracetamol for lower third molar extractions under general anaesthesia: is oral administration inferior? Br J Anaesth. 2013 Mar;110(3):432-7. doi: 10.1093/bja/aes387. Epub 2012 Dec 6. PMID 23220855